CLINICAL TRIAL: NCT05455905
Title: Voice Biomarkers Predictive of Depression and Anxiety: An Observational Study
Brief Title: Voice Biomarkers Predictive of Depression and Anxiety
Status: Completed | Type: Observational
Sponsor: Kintsugi Mindful Wellness, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021/08/25
Record Dates: First submitted 2022-06-29; First posted 2022-07-13 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Depression, Anxiety; Healthy; Mental Health Wellness 1
Keywords: mental health; depression; anxiety; Artificial Intelligence
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main Study Cohort: A web-based audio recording tool will be used to record voice sample answering the prompt, "How are you feeling today?" Participants are asked to speak for 1-minute. Following the recording, participants are asked to complete the Patient Health Questionnaire-9 and Generalized Anxiety Disorder-7 questions.
  Interventions: Diagnostic Test: Patient Health Questionnaire-9; Diagnostic Test: Generalized Anxiety Disorder-7
- Selected Self-Reported Depression Cohort: The Researcher will review Patient Health Questionnaire-9 scores of all the participants and select the subset that self-reported a scored greater than 20, on a scale from 0 to 27. Participants will be approached via email to complete an additional administration of the Patient Health Questionnaire-9 and Generalized Anxiety Disorder-7 questionnaires and be offered resources for depression and anxiety and how to set up an appointment with a mental health professional.
  Interventions: Diagnostic Test: Patient Health Questionnaire-9; Diagnostic Test: Generalized Anxiety Disorder-7; Diagnostic Test: Hamilton Depression Rating Scale; Diagnostic Test: Hamilton Anxiety Rating Scale

INTERVENTIONS:
Diagnostic Test: Patient Health Questionnaire-9 — The Patient Health Questionnaire-9 is a nine question self-administered examination in which the patient indicates how often they have experienced different feelings and sensations in the past two weeks. The Patient Health Questionnaire-9 is scored from 0 to 27 where higher scores are associated with more severe depression.
  Other Names: PHQ-9
Diagnostic Test: Generalized Anxiety Disorder-7 — The Generalized Anxiety Disorder-7 is a seven question self-administered examination in which the patient indicates how often they have experienced different feelings and sensations in the past two weeks. The Generalized Anxiety Disorder-7 is scored from 0 to 21 where higher scores are associated with more severe anxiety.
  Other Names: GAD-7
Diagnostic Test: Hamilton Depression Rating Scale — The Hamilton Depression Rating Scale is administered by a mental health profession and includes twenty-one questions asking about how the participant has been feeling in the past week. The Hamilton Depression Rating Scale is scored from 0 to 45 where higher scores are associated with more severe depression.
  Other Names: HDRS; HAM-D
  Groups: Selected Self-Reported Depression Cohort
Diagnostic Test: Hamilton Anxiety Rating Scale — The Hamilton Anxiety Rating Scale is administered by a mental health profession and includes fourteen questions asking about how the participant has been feeling in the past week. The Hamilton Anxiety Rating Scale is scored from 0 to 56 where higher scores are associated with more severe anxiety.
  Other Names: HARS; HAM-A
  Groups: Selected Self-Reported Depression Cohort

SUMMARY:
The objective of this study is to collect data to improve the sensitivity and specificity of Kintsugi Voice's (formerly KiVATM) predictions on audio files. A web-based audio recording tool will be used to record voice sample and ask participants the PHQ-9 and GAD-7 questions. A voluntary subset of participants will then be assessed by mental health professionals with the Hamilton Depression Rating Scale (HAM-D) and Hamilton Anxiety Rating Scale (HAM-A) scores.

DETAILED DESCRIPTION:
Participants will be recruited via various online mediums to participate in a voluntary observational study. Completing the consent and survey on their smart-phone, tablet, or computer, the participant will be asked to provide a 1-minute response to an audio prompt "How was your day?" After recording their response, the participant will be asked to complete the Patient Health Questionnaire-9 and Generalized Anxiety Disorder-7 measures independently.

In a second voluntary phase of the study, participants who indicated a score higher than 20, will be contacted by the research team via email to determine if they are interested in a voluntary follow-up to their initial study participation. Participants who would like to take part in the additional survey will complete additional voice recording responses to prompts and complete the Patient History Questionnaire and Generalized Anxiety Disorder-7. These participants will be contacted by a Mental Health Professional to discuss seeking mental health resources and clinicians, as well as, complete the Hamilton Depression Rating Scale and Hamilton Anxiety Rating Scale via the telephone.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and or females over the age of 18 at the time of informed consent. Adults with a known history of depression and/or anxiety and adults without a known history of depression and/or anxiety will be included in this study.
* Access to a laptop, smart-phone or tablet with a functioning microphone
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Fluency in English

Exclusion Criteria:

* Visual impairment that would make it difficult for the participant to see the web-based survey
* Motor impairment that would make it difficult for the participant to use the web-based survey

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include males and females fluent in English over the age of 18 in the United States and Canada. Participants both with and without a personal history of depression and/or anxiety are eligible to participate in the study. Participants will require access to a laptop, smartphone, or tablet with a functioning microphone and provide stated willingness to comply with all study procedures and availability for the duration of the study. Participants with a visual or motor impairment that would make it difficult to use the web-based survey will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 19533 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-09-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Through study completion, on average 12months
  Participants will be interviewed by mental health professionals using the clinically validated Hamilton Depression Rating Scale, which has a score range of 0 to 54, where higher scores are associated with higher severity of depression.
Hamilton Anxiety Rating Scale | Through study completion, on average 12 months
  Participants will be interviewed by mental health professionals using the clinically validated Hamilton Anxiety Rating Scale, which has a score range of 0 to 56, where higher scores are associated with higher severity anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hsin Cheng, PhD, Principal Investigator — Kintsugi Mindful Wellness, Inc.
Locations (1):
- Kintsugi Mindful Wellness, Inc., Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Czeisler ME, Lane RI, Petrosky E, Wiley JF, Christensen A, Njai R, Weaver MD, Robbins R, Facer-Childs ER, Barger LK, Czeisler CA, Howard ME, Rajaratnam SMW. Mental Health, Substance Use, and Suicidal Ideation During the COVID-19 Pandemic - United States, June 24-30, 2020. MMWR Morb Mortal Wkly Rep. 2020 Aug 14;69(32):1049-1057. doi: 10.15585/mmwr.mm6932a1. PMID 32790653
- [Background] ADAA. Facts & statistics: Anxiety and Depression Association of America. Retrieved March 05, 2021, from https://adaa.org/about-adaa/press-room/facts-statistics
- [Background] Low DM, Bentley KH, Ghosh SS. Automated assessment of psychiatric disorders using speech: A systematic review. Laryngoscope Investig Otolaryngol. 2020 Jan 31;5(1):96-116. doi: 10.1002/lio2.354. eCollection 2020 Feb. PMID 32128436
- [Background] Mundt JC, Vogel AP, Feltner DE, Lenderking WR. Vocal acoustic biomarkers of depression severity and treatment response. Biol Psychiatry. 2012 Oct 1;72(7):580-7. doi: 10.1016/j.biopsych.2012.03.015. Epub 2012 Apr 26. PMID 22541039
- [Background] Zhang L, Duvvuri R, Chandra KKL, Nguyen T, Ghomi RH. Automated voice biomarkers for depression symptoms using an online cross-sectional data collection initiative. Depress Anxiety. 2020 Jul;37(7):657-669. doi: 10.1002/da.23020. Epub 2020 May 7. PMID 32383335
- [Background] Espinola, CW, Gomes, JC, Pereira, JMS et. al. Detection of major depressive disorder using vocal acoustic analysis and machine learning-an exploratory study. Res. Biomed. Eng. 2021; 37: 53-64.
- [Background] Wang J, Zhang L, Liu T, Pan W, Hu B, Zhu T. Acoustic differences between healthy and depressed people: a cross-situation study. BMC Psychiatry. 2019 Oct 15;19(1):300. doi: 10.1186/s12888-019-2300-7. PMID 31615470
- [Background] He L, Cao C. Automated depression analysis using convolutional neural networks from speech. J Biomed Inform. 2018 Jul;83:103-111. doi: 10.1016/j.jbi.2018.05.007. Epub 2018 May 29. PMID 29852317
- [Background] Ozkanca Y, Ozturk MG, Ekmekci MN, Atkins DC, Demiroglu C, Ghomi RH. Depression Screening from Voice Samples of Patients Affected by Parkinson's Disease. Digit Biomark. 2019 May-Aug;3(2):72-82. doi: 10.1159/000500354. Epub 2019 Jun 12. PMID 31872172
- [Background] Yi H, Smiljanic R, Chandrasekaran B. The Effect of Talker and Listener Depressive Symptoms on Speech Intelligibility. J Speech Lang Hear Res. 2019 Nov 18;62(12):4269-4281. doi: 10.1044/2019_JSLHR-S-19-0112. Print 2019 Dec 18. PMID 31738862
- [Background] Stassen HH, Bomben G, Gunther E. Speech characteristics in depression. Psychopathology. 1991;24(2):88-105. doi: 10.1159/000284700. PMID 1886971
- [Background] Taguchi T, Tachikawa H, Nemoto K, Suzuki M, Nagano T, Tachibana R, Nishimura M, Arai T. Major depressive disorder discrimination using vocal acoustic features. J Affect Disord. 2018 Jan 1;225:214-220. doi: 10.1016/j.jad.2017.08.038. Epub 2017 Aug 16. PMID 28841483
- [Background] Low LS, Maddage NC, Lech M, Sheeber LB, Allen NB. Detection of clinical depression in adolescents' speech during family interactions. IEEE Trans Biomed Eng. 2011 Mar;58(3):574-86. doi: 10.1109/TBME.2010.2091640. Epub 2010 Nov 11. PMID 21075715
- [Background] Tuka A, Mohammad G, and James G. Detecting Depression with Audio/Text Sequence Modeling of Interviews. Interspeech. 2018; 2522.
- [Background] Pan W, Flint J, Shenhav L, Liu T, Liu M, Hu B, Zhu T. Re-examining the robustness of voice features in predicting depression: Compared with baseline of confounders. PLoS One. 2019 Jun 20;14(6):e0218172. doi: 10.1371/journal.pone.0218172. eCollection 2019. PMID 31220113
- [Background] Xu, M, Duan, LY, Cai, J, Chia, LT, Xu, C, & Tian, Q. HMM-based audio keyword generation. In Pacific-Rim Conference on Multimedia. 2004; November: 566-574. Springer, Berlin, Heidelberg.
- [Background] Aizawa IK, Nakamura Y, Satoh S, et. al. Advances in Multimedia Information Processing - PCM 2004: 5th Pacific Rim Conference on Multimedia. Springer. ISBN 978-3-540-23985-7.
- [Background] Crockford, D. (2001, April). Introducing JSON. JavaScript Object Notation. https://www.json.org/json-en.html
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Trajkovic G, Starcevic V, Latas M, Lestarevic M, Ille T, Bukumiric Z, Marinkovic J. Reliability of the Hamilton Rating Scale for Depression: a meta-analysis over a period of 49 years. Psychiatry Res. 2011 Aug 30;189(1):1-9. doi: 10.1016/j.psychres.2010.12.007. Epub 2011 Jan 26. PMID 21276619
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508

DOCUMENTS (2):
  • Study Protocol (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT05455905/Prot_000.pdf
  • Informed Consent Form (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT05455905/ICF_001.pdf